CLINICAL TRIAL: NCT04627948
Title: STHLM3 AS NorDCaP - a Followup Study of Men on Active Surveillance of Prostate Cancer
Acronym: NorDCaP AS
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Helse Stavanger HF (Other Government); University of Aarhus (Other); Mehiläinen, Finland (Unknown); Capio Sankt Görans Hospital (Other)
Responsible Party: Principal Investigator, Anna Lantz, MD PhD Principal Investigator, Karolinska Institutet
Other Study IDs: 2019-02020
Record Dates: First submitted 2020-11-05; First posted 2020-11-13 (Actual); Last update posted 2025-01-21 (Actual); Status verified 2022-12

CONDITIONS: Prostate Cancer
Keywords: Active Surveillance
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Stockholm3 test — Diagnostic test: Stockholm3-test. Men from the study sites, diagnosed with prostate cancer and currently on AS and planned for rebiopsies will be invited to the study.

SUMMARY:
The aim of the STHLM3 AS NorDCaP study is to evaluate the Stockholm3 test in an active surveillance cohort to predict upgrading on rebiopsy. The study follows a paired design, evaluating our proposed protocol for follow up men on active surveillance with Stockholm3 versus the standard protocol according to national guidelines with PSA.

DETAILED DESCRIPTION:
STHLM3 AS NorDCaP is a cross-sectional multi-center study, evaluating the predictive value of Stockholm3 test in a prostate cancer cohort on AS for upgrading on rebiopsy. Men from the study sites, diagnosed with prostate cancer and currently on AS and planned for rebiopsies will be invited to the study. Eligible individuals have to be alive without any severe comorbidity and without a history of initiating treatment; surgery, radiation, hormone therapy or chemotherapy. To avoid the need for additional investigations, sampling will be synchronized with timing for planned follow-up within the AS program for each individual.

At baseline blood will be drawn for Stockholm3 analyses. The patient will be asked to fill out an informed consent. For each man the following data will be collected: Stockholm3 Risk Score, Stockholm3 Prostate Volume cut-off, total PSA, DRE status, MRI results (PI-RADS, optional, only if MRI is conducted within 3 months before biopsy), prostate volume, biopsy results (ISUP, cancer length, number of positive cores, total number of cores and stage).

Main outcome measurement will be number of upgrading, i.e. number of detected ISUP ≥ 2 cancers.

ELIGIBILITY:
Inclusion Criteria:

* Men diagnosed with low-risk PC and currently on AS and planned for follow-up with systematic and/or fusion biopsies as following standard of care.

Exclusion Criteria:

* History of treatment for prostate cancer; surgery, radiation, chemotherapy or hormonal treatment.
* Severe illnesses such as metastatic cancers, severe cardio-vascular disease or dementia

Ages: 40 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men diagnosed with low-risk PC, currently on AS and planned for follow-up with biopsies from the different inclusion sites will be invited to the study. Potential participants will be invited to the study by their urologist at their yearly follow up.
Sampling Method: Non-Probability Sample
Enrollment: 199 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Validate if the Stockholm3 test can be used in an AS cohort to predict upgrading | Through study completion, an average of 1 year
  Number of ISUP ≥ 2 prostate cancer

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska Institutet, Stockholm, Solna, Sweden

IPD SHARING:
Plan to Share IPD: No
Information obtained in the study will be collected in one database. The purpose of the database is to collect study data in a proper and safe way for a long time. All information about the participants will be treated with utmost confidentiality and with strong safeguards to preserve their anonymity. All data and test results will be treated to prevent unauthorized access to them. The samples will get a unique code so that outsiders cannot identify them. The participants' samples are treated in accordance with the National Biobank Act and other relevant laws.
  Everyone who works with STHLM3 AS NorDCaP are under confidentiality agreements. Results from the study are presented only as statistics in which individual answers cannot be traced.
  Treatment of the personal data is in accordance with GDPR and other relevant national laws.